CLINICAL TRIAL: NCT06868589
Title: Randomized Clinical Trial of Methadone and Ketamine for Pain Management During Deceased Donor Liver Transplant
Brief Title: Reducing Pain With Methadone and Ketamine in Liver Transplant
Acronym: RELIEF-LT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Lahey Clinic (Other)
Responsible Party: Principal Investigator, Ryan Nazemian, Staff Anesthesiologist: Division of Transplant, Director: Transplant Anesthesia Fellowship, Co-Director: Anesthesia Informatics, Lahey Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20243140
Record Dates: First submitted 2025-03-01; First posted 2025-03-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-06

CONDITIONS: Liver Transplantation
Keywords: Liver Transplantation; Deceased Donor Liver Transplant; Postoperative Pain; Methadone; Ketamine; Perioperative Analgesia; Anesthesiology; Acute Pain; Transplant Surgery; Opioids
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Methadone; Ketamine; Hydromorphone; Fentanyl

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either intervention or standard of care group at the ratio of 1:1
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants won't be aware of the study arm and treatments they receive. The statistician will be masked on the treatment group during final study analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- M+K group (Experimental): Participants in this arm will receive the intervention with methadone and ketamine
  Interventions: Drug: Methadone; Drug: ketamine
- SOC group (Active Comparator): Participants in this arm will receive the standard of care with combination of hydromorphone and fentanyl
  Interventions: Drug: Hydromorphone; Drug: fentanyl

INTERVENTIONS:
Drug: Methadone — Participants in this group will receive one bolus dose of intravenous Methadone and Ketamine at the start of operation
  Arms: M+K group
Drug: ketamine — Participants in this group will receive one bolus dose of intravenous Methadone and Ketamine at the start of operation
  Arms: M+K group
Drug: Hydromorphone — Participants in this group will receive standard of care for pain with either intravenous fentanyl and/or hydromorphone boluses during the procedure
  Arms: SOC group
Drug: fentanyl — Participants in this group will receive standard of care for pain with either intravenous fentanyl and/or hydromorphone boluses during the procedure
  Arms: SOC group

SUMMARY:
The goal of this clinical trial is to learn if using methadone and ketamine during an adult deceased donor liver transplant can help decrease pain after surgery.

The main questions it aims to answer are:

* What impact does using methadone and ketamine during a deceased donor liver transplant have on pain after surgery?
* Does the use of methadone and ketamine also have an impact on mental confusion (delirium) after surgery?

Researchers will compare the use of methadone and ketamine to standard of care to see if the two drugs work to decrease pain and impact delirium after liver transplant.

Participants will:

* Receive either methadone and ketamine or standard of care during their deceased donor liver transplant.
* Allow researchers to follow medical care throughout inpatient stay.

DETAILED DESCRIPTION:
Pain control following liver transplantation (LT) has been the subject of interest of many research projects due to invasive nature of the procedure, significant comorbidities of recipients, effect of hepatic metabolism on many common pain medications and difficulties in performing some neuraxial and regional techniques given patient coagulopathy. Some newer regional nerve blocks such as External Oblique Intercostal (EOI) block has also been successfully utilized in pain management of patients undergoing liver resections but their utilization in perioperative setting for high-MELD patients and after-hour operations are limited. Methadone and ketamine are well-known drugs that have been recently emerged as components of new pain management pathways in many open surgeries due to their availability, cost, well-known metabolism, good safety profile and prolonged effects. Evidence has emerged that their use is associated with decreased likelihood of development of chronic pain and need for long term opioids. The combination of methadone and ketamine has been shown to be superior to opioids alone due to synergistic effect on N-methyl-d-aspartate and μ-opioid receptors. But these medications have not been extensively studied in LT recipients except for a few case reports and small studies. Current standards of care for intraoperative pain management during LT are systemic short and medium long-acting opioids such as fentanyl and hydromorphone which both have numerous concerns such as respiratory depression and opioid dependency. The aim of this study is to prospectively evaluate the effect of intraoperative methadone and ketamine administration on postoperative pain in liver transplant recipients. These drugs have been safely used during liver transplantation at LHMC and other centers and showed to be effective and safe, but the exact dosing and timing of administration requires further studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age at the time of LT.
* Undergoing LT from a deceased donor.
* Written informed consent obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion criteria:

* Living donor liver transplantation (LDLT).
* Split liver transplantation (isolated right or left lobe).
* Acute liver failure (ALF) as the indication for LT.
* Repeat (redo) liver transplant
* Simultaneous liver and kidney transplant (SLK)
* Sedation or high vasopressor use.
* Subject is intubated and/or mechanically ventilated prior to entering the operating room for LT.
* Severe Hepatic encephalopathy
* History of psychiatric disorders such as schizophrenia or bipolar mood disorders
* History of chronic opioid use, substance abuse or opioid maintenance therapies
* Any history of allergic reaction to any of the study drugs History of Brugadda, prolonged QT syndrome or QTc in preoperative setting
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data
* Prisoner
* Pregnant person
* Operational Exclusion Criterion: Subjects will not be enrolled if study personnel required for protocol execution (e.g., study investigator, research staff or pharmacy staff) are unavailable at the time of transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | 8, 16, 24, 32, 40 and 48hours post-surgery finish
  postoperative opioid consumption (measured as morphine milligram equivalents ((MME)) 48 hours after surgery
Postoperative Pain | 8, 16, 24, 32, 40 and 48hours post-surgery finish
  Subjective postoperative pain scores measured as 0-10 (10 being the worst pain)

SECONDARY OUTCOMES:
Length of stay in intensive care unit | Post surgery finish until discharge from intensive care unit, or date of death from any cause, whichever came first, assessed up to 30 days
  Duration of length of stay in intensive care unit in hours
Length of stay in hospital | Post surgery finish until discharge from hospital, or date of death from any cause, whichever came first, assessed up to 30 days
  Duration of length of stay in the hospital in days
Delirium | Post surgery finish until discharge from intensive care unit, or date of death from any cause, whichever came first, assessed up to 30 days
  Incidence of postoperative delirium measured by standard CAM-ICU scores, ICD-10 diagnosis of delirium, any use of anti-agitation medication such as haloperidol, dexmedetomidine or seroquel
Respiratory complications | Post surgery finish until discharge from intensive care unit, or date of death from any cause, whichever came first, assessed up to 30 days
  Any significant respiratory complications such as re-intubation, need for invasive ventilation such as BIPAP or CPAP
Narcotics reversal agent | Post surgery finish until discharge from intensive care unit, or date of death from any cause, whichever came first, assessed up to 30 days
  Any need for narcotics reversal agents such as Naloxone after administration of study drugs
Postoperative adjunct pain modalities | Post surgery finish until discharge from intensive care unit, or date of death from any cause, whichever came first, assessed up to 30 days
  Incidence of usage of any additional pain modalities such as nerve blocks, neuraxial anesthesia, non-narcotic pain medications such as additional ketamine dose, ketorolac, methocarbamol, ketorolac, etc
Correlation Between Study Drug Exposure and Early Post-Transplant Laboratory Markers of Liver Dysfunction | Immediate to 24hrs post surgery finish
  Unit of measure: Correlation coefficient (r) describing the association between study drug exposure and postoperative laboratory markers of liver dysfunction during the first 24hrs post surgery.
  Independent variables (study drug exposure):
  * Randomized study drug assignment (e.g., ketamine vs methadone vs standard of care)
  * Total intraoperative dose of each study drug (total mg)
  Dependent variables (markers of postoperative liver dysfunction):
  Correlation coefficients will be calculated between study drug exposure and the following laboratory values measured during first postoperative days :
  * Peak alanine aminotransferase (ALT), IU/L
  * Peak aspartate aminotransferase (AST), IU/L
  * Peak total bilirubin, mg/dL
  * Peak international normalized ratio (INR)
Correlation Between Donor and Surgical Factors and Postoperative Opioid Use (MME) | From the end of surgery through 48hr post surgery
  Unit of measure: Correlation coefficient (r) describing the association between each donor/surgical factor and total postoperative opioid consumption (MME) during postoperative days 0-2. Total MME will be calculated by converting all administered opioids into morphine milligram equivalents using standard conversion factors.
  Factors assessed (independent variables):
  * Donor age (years)
  * Donation type (donation after brain death vs donation after circulatory death)
  * Use of normothermic machine perfusion (yes/no)
  * Cold ischemia time (hours)
  * Warm ischemia time (minutes)
  * Surgical technique characteristics (e.g., piggyback vs caval replacement approach, vascular anastomosis techniques, use of veno-venous bypass), coded as categorical variables

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Nazemian, MD, PhD, Principal Investigator — Lahey Hospital and Medical Center, Department of Anesthesiology, Perioperative and Pain Medicine
Locations (1):
- Lahey Hospital and Medical Center, Burlington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Sensitive transplant data will not be shared for patients privacy